CLINICAL TRIAL: NCT02550249
Title: Phase II Study of Neoadjuvant Nivolumab in Patients With Glioblastoma Multiforme
Brief Title: Neoadjuvant Nivolumab in Glioblastoma
Acronym: Neo-nivo
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Clinica Universidad de Navarra, Universidad de Navarra (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Neo-nivo
Record Dates: First submitted 2015-07-16; First posted 2015-09-15 (Estimated); Last update posted 2017-04-11 (Actual); Status verified 2015-07

CONDITIONS: Glioblastoma Multiforme
MeSH Terms: conditions — Glioblastoma | interventions — Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Nivolumab (Experimental): Nivolumab 3 mg every 2 weeks
  Interventions: Drug: Nivolumab

INTERVENTIONS:
Drug: Nivolumab — Intravenous administration of nivolumab
  Other Names: Opdivo

SUMMARY:
Neoadjuvant nivolumab will be administered to patients with primary and recurrent glioblastoma multiforme that require surgery. Nivolumab will be continued following surgery.

DETAILED DESCRIPTION:
Neoadjuvant nivolumab will be administered to patients with primary and recurrent glioblastoma multiforme that require surgery. Nivolumab will be continued following surgery until toxicity or progression.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent.
* Patients must be willing and able to comply with scheduled visits, treatment schedule, laboratory testing and other requirements of the study.
* Patients with GBM that are candidates to primary or salvage resection surgery, according to the following criteria:
* Patients may have received previous treatments for GBM. There is no limit on previous treatment lines, as long as the other inclusion criteria are met.
* Patients in whom surgery can be safely delayed for a minimum period of 2 weeks following the administration of the first dose of nivolumab, in the opinion of the investigator.
* Eastern Cancer Oncology Group (ECOG) performance status of 0-1. Patients with ECOG>1 due to neurological symptoms considered to be reversible following surgery, according to investigator´s criteria will be eligible
* Life expectancy >12 weeks.
* Adequate organ function defined by:

  1. Bone Marrow Reserve: white blood cells (WBC): ≥2000/ mm3 absolute neutrophil count (ANC) ≥1500x 109/L; platelet count ≥100000/ mm3 100 x 109/L; hemoglobin ≥9.0 g/dL).
  2. Hepatic: bilirubin <1.5 times the upper limit of normality (ULN), AST and ALT <3.0 × ULN (BR< 3 x ULN for patients with Gilbert´s Syndrome).
  3. Renal: creatinine < 1.5 x ULN or estimated creatinine clearance > 40 ml/min, using the Cockcroft-Gault formula.

Exclusion Criteria:

* Presence of extracranial disease.
* Any serious or uncontrolled medical disorder that, in the opinion of the investigator, may increase the risk associated with study participation or study drug administration, impair the ability of the subject to receive the planned therapy (including brain surgery), or interfere with the interpretation of study results.
* Subjects with active, known or suspected autoimmune disease. Subjects with vitiligo, type I diabetes mellitus, residual hypothyroidism due to autoimmune condition only requiring hormone replacement, psoriasis not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger are permitted to enroll.
* Previous treatment with a PD-1, PDL1 or CTLA-4 targeted therapy
* Treatment with any anti-cancer drug or radiation therapy within the last 14 days. A shorter interval can be approved by the principal investigator, if deemed appropriate.
* Patients should be excluded if they have a condition requiring systemic treatment with either corticosteroids (>10 mg daily prednisone equivalents), with the exception of control of cerebral edema, or other immunosuppressive medications within 14 days of study drug administration. Inhaled or topical steroids and adrenal replacement doses > 10 mg daily prednisone equivalents are permitted in the absence of active autoimmune disease.
* Pregnant or breastfeeding patients.
* Known history of testing positive for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS). Routine testing is not required.
* Positive tests for hepatitis B virus surface antigen (HBV sAg) or hepatitis C virus ribonucleic acid (HCV RNA) indicating active or chronic infection.
* History of allergy to study drug components or of severe hypersensitivity reactions to any monoclonal antibodies.
* Prisoners or subjects who are involuntarily incarcerated or who are compulsorily detained for treatment of either a psychiatric or physical (eg, infectious disease) illness.
* Subjects unable (due to existent medical condition, e.g, pacemaker or implantable cardioverter defibrillator device) or unwilling to have a head contrast enhanced MRI and/or a CT scan of the brain.
* Concomitant or prior malignancy that, in the opinion of the investigator contraindicates GBM surgery or can interfere with the results of the study, in the opinion of the investigator.
* Known drug or alcohol abuse.

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2015-06; Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Changes in percentage and level of expression of Programmed Death-Ligand 1 (PD-L1) by tumor cells and lymphocytes, assessed at baseline and following neoadjuvant nivolumab in Glioblastoma multiforme (GBM). | 1 neoadjuvant cycle followed by surgery (4 weeks). Evaluation will be performed at baseline and after the neoadjuvant cycle
  We will assess levels of expression of Programmed Death-Ligand 1 (PD-L1) by tumor cells and lymphocytes at baseline and following neoadjuvant nivolumab in Glioblastoma multiforme (GBM). The specific outcome will be the changes in these levels.

SECONDARY OUTCOMES:
Efficacy: response rate assessed by Response Assessment in Neuro-Oncology (RANO) criteria | 1 neoadjuvant cycle followed by surgery (4 weeks)
Safety: toxicity assessed by Common Toxicity Criteria (CTC) version 4 | 1 neoadjuvant cycle followed by surgery (4 weeks)

CONTACTS AND LOCATIONS:
Overall Officials: Ignacio Melero, MD, PhD, Principal Investigator — Clinica Universidad de Navarra
Locations (1):
- Clinica Universidad de Navarra, Pamplona, Navarre, Spain